CLINICAL TRIAL: NCT03398993
Title: Comparative Study of Pregnancy Rate After Endometrial Injury in Couples With Unexplained Infertility
Brief Title: Effect of Endometrial Injury in Couples With Unexplained Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Clomiphene; Chorionic Gonadotropin; hMG-IBSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scratch group (Active Comparator): Induction of ovulation will be done by clomophine citrate from 3rd day of cycle till 7th day of cycle and HMG 75IU (MerionaL) given from 6th day of cycle till 8th of cycle once daily. folliculometry done regularly during induction of ovulation till dominant follicle reached 18_20mm in size.
  Then endometrial injury performed in pre ovulatory day by a thin pipelle (a fine, flexible, sterile, plastic tube) The procedure was carried out in preovulatory day (known when dominant follicle reached 18_20 mm in diameter), usually, done around day 14-day of the cycle
  Interventions: Drug: Clomiphene Citrate; Drug: Human chorionic gonadotropin; Device: Endometrial scratch
- Non scratch group (Active Comparator): They will receive the same induction of ovulation as first group but without performing endometrial injury in preovulatory day
  Interventions: Drug: Clomiphene Citrate; Drug: Human chorionic gonadotropin

INTERVENTIONS:
Drug: Clomiphene Citrate — 50 mg twice daily from3rd day of cycle till 7th day of cycle
  Other Names: clomid
Drug: Human chorionic gonadotropin — 75 IU dail;y from 6th day of cycle till 8th of cycle once daily
  Other Names: MerionaL
Device: Endometrial scratch — The procedure was carried out in preovulatory day (known when dominant follicle reached 18_20 mm in diameter), usually, done around day 14-day of the cycle.
  In the theatre, Patients put in a lithotomy position, sterilization was performed with the presence of good source of light., the procedure was carried out using a thin pipelle tube as follow :- A cuscoe's speculum was inserted into the vagina in order to visualize the cervix.
  Cervix was grasped by vollselum upwards backwards, then pipelle tube passed through the cervix and uterine cavity, then moved up and down to make a single induced scratch two times in the lining endometrium of posterior wall of uterus.
  The procedure took approximately 15minutes to complete
  Arms: Scratch group

SUMMARY:
100 patient of unexplained infertility recruited and divided into two groups for the study group (50) endometrial scratching done in preovulatory period after controlled ovarian stimulation by clomiphene citrate , then followed and compared to control group for 6 months to asses pregnancy rate

DETAILED DESCRIPTION:
Induction of ovulation was done by clomophine citrate (selective estrogen modulator of triphenylethylene group, produced by( Sanafi Aventis company) from 3rd day of cycle till 7th day of cycle and HMG 75IU (MerionaL) produced by IBSA ( Institute biochimique SA) given from 6th day of cycle till 8th of cycle once daily. folliculometry done regularly during induction of ovulation till dominant follicle reached 18_20mm in size.

Then endometrial injury performed in pre ovulatory day by a thin pipelle (a fine, flexible, sterile, plastic tube) produced by Jiangsu Guard King Medical Equipment Co.

The procedure was carried out in preovulatory day (known when dominant follicle reached 18_20 mm in diameter), usually, done around day 14-day of the cycle.

In the theatre, Patients put in a lithotomy position, sterilization was performed with the presence of good source of light., the procedure was carried out using a thin pipelle tube as follow :- A cuscoe's speculum was inserted into the vagina in order to visualize the cervix.

Cervix was grasped by vollselum upwards backwards, then pipelle tube passed through the cervix and uterine cavity, then moved up and down to make a single induced scratch two times in the lining endometrium of posterior wall of uterus.

The procedure took approximately 15minutes to complete. It was uncomfortable or painful in some circumstances and that bleeding after the procedure happened in many cases. Post procedure antibiotics were given.

Couples were advised to practice timed sexual intercourse for next 6months and couples in both groups were asked to phone a contact Person whenever there was a missed period. The patients followed up for six months for detecion of the biochemical pregnancy if occurred.

2- Control group (50patients) :- They received the same induction of ovulation as first group but without performing endometrial injury in preovulatory day.

We wait till time of period if missed period achieved serum pregnancy test done after one week of missed period .

All women followed for 6 months after treatment. Comparative study was done for both groups and results presented in tables and statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility ( 1ry & 2ndry infertility) : *

  * Normal hormonal profile of infertile woman.
  * Normal hystrosalpingogram.
  * Normal laparoscopy.
  * Normal investigation of the cervical factor
  * Fertile semen analysis (according to world health organization criteria 2015).

Exclusion Criteria:

* • Infertile semen analysis.

  * Abnormal HSG.
  * Abnormal laparoscopic findings.
  * Disturbed hormonal profile.
  * Evidence of cervical factor.
  * Known genetic disorder
  * Known autoimmune disease

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after missed period
  intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided